CLINICAL TRIAL: NCT06799364
Title: A Randomised, Controlled, Double-blind, Three Parallel Groups, Multi-centre Study to Assess the Bifidobacterium Diversity After 28-days Consumption of Fermented Dairy Products With Three Bifidobacterium Strains With or Without Galacto-oligosaccharides Compared to Yoghurt in 45 to 60-year-old Healthy Subjects
Brief Title: Fermented Dairy Product and Bifidobacterium Diversity (ThreeBees)
Acronym: ThreeB (TB)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 23REX0060156
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: A03 - Digestive System; B03 - Bacteria
Keywords: Gut microbiota; Fibre; Yoghurt; Bifidobacteria diversity; Galacto-oligosaccharides
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral administration of experimental product A (Experimental): Test product A: fermented dairy product containing Bifidobacterium strains
  Interventions: Other: 28-days consumption of Product A in 45 to 60-year-old healthy subjects.
- Oral administration of experimental product B (Experimental): Test product B: product A with galacto-oligosaccharides (GOS)
  Interventions: Other: 28-days consumption of Product B in 45 to 60-year-old healthy subjects.
- Oral administration of Control product (Placebo Comparator): Control product: commercially available yoghurt
  Interventions: Other: 28-days consumption of Control product in 45 to 60-year-old healthy subjects.

INTERVENTIONS:
Other: 28-days consumption of Product A in 45 to 60-year-old healthy subjects. — 48 healthy volunteers will consume Product A twice per day during 28 consecutive days.
  Arms: Oral administration of experimental product A
Other: 28-days consumption of Product B in 45 to 60-year-old healthy subjects. — 48 healthy volunteers will consume Product B twice per day during 28 consecutive days.
  Arms: Oral administration of experimental product B
Other: 28-days consumption of Control product in 45 to 60-year-old healthy subjects. — 48 healthy volunteers will consume Control product twice per day during 28 consecutive days.
  Arms: Oral administration of Control product

SUMMARY:
Bifidobacterium strains with potential health benefits can contribute to the gastrointestinal wellbeing. However, the ability of these strains to survive gastro-intestinal tract stress and their impact on gut microbiome remains to be clarified. Moreover, prebiotic fibres, such as galacto-oligosaccharides (GOS) can promote the proliferation of Bifidobacteria. This is why the current study aims to assess the impact of Bifidobacteria consumption on human gut microbiome with or without GOS compared to control product.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged between 45 and 60 years old.
2. BMI between 18.5 kg/m2 and 30 kg/m2.
3. Subjects who are overtly healthy as determined by the investigator.
4. Willing and/or able to:

   * Speak and read in French,
   * Collect, store and transport their faecal samples themselves,
   * Consume the study products twice per day for 28 consecutive days and not to consume any fermented dairy products during the entire study (other than the study products) as well as any probiotic, prebiotic or synbiotic supplements during the entire study.
   * Complete the electronic Patient Reported Outcomes (ePRO) using their own digital device having access to internet.
5. Willing to limit alcohol consumption and not to smoke or consume any soft or hard drug during the study.
6. Having access to adequate space to store the investigational products in their own fridge at home.
7. Having regular bowel movements.
8. Signed written informed consent by the participant.
9. Female subjects must either be postmenopausal for at least 12 months or have undergone specific surgical procedures resulting in sterility or they are using one of the medically approved contraceptive methods.
10. Subject is covered by French health insurance.
11. Subject agrees to be registered in the national database of subjects participating in clinical research.

Exclusion Criteria:

1. Any ongoing metabolic disease, hypertension, inflammatory disease, allergic conditions requiring chronic systemic medication, psychiatric disorder, gastrointestinal disorder, chronic pain, or neurological disorder diagnosed by a physician.
2. Known allergy or intolerance to any ingredients or potential allergens.
3. Pregnancy or breast-feeding at the screening visit or plan for pregnancy during the study.
4. Any antecedents or plan for digestive or dental surgery, general anaesthesia or any participation in another study with investigational or marketed products potentially affecting the gut microbiota.
5. Unable (or unwilling) to adhere to protocol requirements (based on investigator's judgement).
6. Subject with a special diet at the screening visit, or plan for such diet during the study.
7. Major changes in subject's dietary habits ≤ 4 weeks before the screening visit or plan for such major changes during the study including change in vitamin or mineral supplements use, but except for dietary restrictions related to the study.
8. Enhanced diet together with intense physical activity ≤ 4 weeks before the screening visit, plan for such a diet and training during the study, or plan for major changes in physical activity during the study.
9. Use ≤ 8 weeks before the screening visit or plan of use during the study of systemic medication that can affect the gastrointestinal function or plan of use during the study (if needed, incidental use of ≤ 4 tablets of paracetamol, non-steroidal anti-inflammatory drugs (NSAIDs) or aspirin per 2-week period is allowed).
10. Subject with excessive alcohol consumption, active smoker or quit active smoking less than 5 years ago before the screening visit. Not regularly smoking is allowed.
11. Drug abuse based on investigator's judgement.
12. Living in the same home as others already participating in the study and to concomitantly receive some study products.
13. Subject under guardianship, curatorship, person under judicial protection, family empowerment or future protection mandate.
14. Employees, family members or other relatives of employees of the participating centre or of Danone Global Research & Innovation Center.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 182 (Actual)
Dates: Start 2025-02-21 (Actual); Primary Completion 2025-12-22 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
The primary outcome parameter in this study is the change from baseline after 28-days product consumption of the number of distinct Bifidobacterium species. | After 28 days of study product consumption

SECONDARY OUTCOMES:
The changes from baseline after 28-days product consumption in detection and quantification of viable bacteria (i.e. with intact cell membrane) for the Bifidobacterium strains. | After 28 days of study product consumption
The change from baseline after 28-days product consumption of Bifidobacterium diversity indices. | After 28 days of study product consumption

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CEN, Dijon
  - Biofortis, Paris
  - Biofortis, Saint-Herblain

IPD SHARING:
Plan to Share IPD: No